CLINICAL TRIAL: NCT00867022
Title: Autonomic Nervous Activity in Women With Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Risto Kaaja, Helsinki University Hospital
Other Study IDs: GESTSYMPIS
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2009-03-23 (Estimated); Status verified 2009-03

CONDITIONS: Gestational Diabetes
Keywords: Inflammatory factors; Coagulation factors; Sympathetic activity
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Women with gestational diabetes
- 2: Pregnant women without gestational daibetes
- 3: Women with gestational diabetes and hypertension
- 4: Non pregnant women

SUMMARY:
Through complex hormonal pathways, insulin resistance can lead to the activation of the sympathetic nervous system, and vice versa. Schobel et al. showed that in PE patients, mus-cle sympathetic nerve activity (MSNA) is increased compared with normotensive pregnant and non-pregnant women. Studies assessing heart-rate variability and plasma noradrenalin concentrations also suggest increased sympathetic activity in PE. It has been hypothesized that sympathetic over-activity is a precursor of PE, normally compensated for by vasodilating mechanisms, but resulting in PE when the mechanisms fail. In addition to sympathetic activity, various markers of inflamma-tion are also associated with reduced insulin sensitivity, suggesting that chronic sub-clinical inflamma-tion could be part of the insulin resistance syndrome. The role of sympathetic over-activity and inflammatory markers in gestational diabetes has not been investigated

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gestational diabetes (OGTT) with or without BP > 140/90.
* Pregnant control with normal OGTT-

Exclusion Criteria:

* Smoking
* Uncontrolled hypertension
* Diabetes
* Medication affecting sympathetic activity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Gestational diabetic women having or not hypertension with two control groups, one pregnant on non-pregnant. All the women are studied during night time to study the arousal of the sympathetic activity in the early morning hours
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2004-08; Primary Completion 2007-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Serum Noradrenalin level

SECONDARY OUTCOMES:
Heart rate variability: LF, VLF, HF

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstet and Gyn, Helsinki University Hospital, Helsinki, Uusimaa, Finland